CLINICAL TRIAL: NCT03822078
Title: A Randomized, Double-blind, Placebo-controlled, Single-dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of AMG 162 Administered Subcutaneously to Japanese Postmenopausal Women
Brief Title: Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Denosumab (AMG 162) in Japanese Postmenopausal Women
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: 20030164
Record Dates: First submitted 2019-01-28; First posted 2019-01-30 (Actual); Results first posted 2019-07-24 (Actual); Last update posted 2019-07-24 (Actual); Status verified 2019-05

CONDITIONS: Osteoporosis
Keywords: Postmenopausal; Denosumab
MeSH Terms: conditions — Osteoporosis | interventions — Denosumab

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Placebo (Placebo Comparator): Participants received a single subcutaneous injection of placebo to denosumab on day 1.
  Interventions: Drug: Placebo
- Denosumab (Experimental): Participants received a single subcutaneous dose of denosumab on day 1. Doses included 0.03, 0.1, 0.3, 1.0, and 3.0 mg/kg.
  Interventions: Biological: Denosumab

INTERVENTIONS:
Drug: Placebo — Administered by subcutaneous injection
  Arms: Placebo
Biological: Denosumab — Administered by subcutaneous injection
  Other Names: AMG 162; Prolia
  Arms: Denosumab

SUMMARY:
The primary objective was to evaluate the safety and tolerability of denosumab (AMG 162) after a single subcutaneous administration in Japanese postmenopausal women.

ELIGIBILITY:
Inclusion Criteria:

* ambulatory women between the ages of 40 and 64 years, inclusive
* postmenopausal, defined as amenorrheic for at least 24 months
* clinically acceptable physical exam
* clinical laboratory tests (complete blood count [CBC], blood chemistries, urinalysis) within normal limits or clinically acceptable to the investigator/sponsor at the time of screening with the exception of aspartate transaminase (AST) and alkaline phosphatase (ALT), which must be < 1.25 times the upper limit of normal, or gamma-glutamyl transpeptidase (GGT), which must be < 1.5 times the upper limit of normal
* normal or clinically acceptable electrocardiogram (ECG) (12-lead reporting ventricular rate and PR, QRS, QT, and QTc intervals)
* body mass index between 17 and 27
* willing to sign an approved informed consent form before any study-specific assessments and oral consultations are performed

Exclusion Criteria:

* administration of medications within 6 months before investigational product administration that are known to effect bone metabolism, including but not limited to the following: calcitonin, parathyroid hormone (or any derivative), supplemental vitamin D (> 1000 IU/day), glucocorticosteroids (inhaled or topical corticosteroids administered more than 2 weeks before the date of informed consent were allowed), anabolic steroids, calcitriol and available analogues, diuretics
* administration of the following medications within 12 months before study drug administration: bisphosphonates, fluoride for osteoporosis
* diagnosed with any condition that affects bone metabolism
* greatly differing levels of physical activity compared with the 6 months before investigational product administration or constant levels of intense physical activities
* routine alcohol intake of ≥ 2 drinks/day, on average, within 6 months of investigational product administration
* known sensitivity to any drugs
* positive test results for hepatitis B surface antigen, hepatitis C virus, human immunodeficiency virus antigen/antibody, syphilis
* receiving or received any investigational drug (or was currently using an investigational device) within 4 months before receiving investigational product
* donated any amount of blood within 16 weeks, or over 400 mL (Note: not 400 mL but 200 mL, for the subjects who were to be enrolled into cohorts 4 or 5) within 1 year of the start day of screening
* subject had previously entered this study
* any other condition that might have reduced the chance of obtaining data (eg, known poor compliance) required by the protocol or that might have compromised the ability to give truly informed consent

Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2003-09-30 (Actual); Primary Completion 2004-12-24 (Actual); Study Completion 2004-12-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kumagai Y, Hasunuma T, Padhi D. A randomized, double-blind, placebo-controlled, single-dose study to evaluate the safety, tolerability, pharmacokinetics and pharmacodynamics of denosumab administered subcutaneously to postmenopausal Japanese women. Bone. 2011 Nov;49(5):1101-7. doi: 10.1016/j.bone.2011.08.007. Epub 2011 Aug 12. PMID 21871589
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at one clinical center in Japan.
Pre-assignment Details: The study consisted of 5 dose cohorts of 8 participants. Within each dose cohort 6 participants were randomly assigned to receive denosumab and 2 participants to receive placebo.
Groups:
- Denosumab 0.03 mg/kg: Participants received a single subcutaneous injection of 0.03 mg/kg denosumab on day 1.
- Denosumab 0.1 mg/kg: Participants received a single subcutaneous injection of 0.1 mg/kg denosumab on day 1.
- Denosumab 0.3 mg/kg: Participants received a single subcutaneous injection of 0.3 mg/kg denosumab on day 1.
- Denosumab 1.0 mg/kg: Participants received a single subcutaneous injection of 1.0 mg/kg denosumab on day 1.
- Denosumab 3.0 mg/kg: Participants received a single subcutaneous injection of 3.0 mg/kg denosumab on day 1.
Period: Overall Study
Arm/Group | Placebo | Denosumab 0.03 mg/kg | Denosumab 0.1 mg/kg | Denosumab 0.3 mg/kg | Denosumab 1.0 mg/kg | Denosumab 3.0 mg/kg
Started | 12 | 6 | 6 | 8 | 7 | 6
Received Study Drug | 10 | 6 | 6 | 6 | 6 | 6
Completed | 10 | 6 | 6 | 6 | 6 | 6
Not Completed | 2 | 0 | 0 | 2 | 1 | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Denosumab 0.03 mg/kg | Denosumab 0.1 mg/kg | Denosumab 0.3 mg/kg | Denosumab 1.0 mg/kg | Denosumab 3.0 mg/kg | Total
Number analyzed (Participants) | 12 | 6 | 6 | 8 | 7 | 6 | 45
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.83 (2.86) | 59.67 (2.34) | 59.50 (3.39) | 58.88 (3.80) | 56.43 (3.95) | 58.67 (2.34) | 58.91 (3.22)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 6 | 6 | 8 | 7 | 6 | 45
  Male | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Japanese | 12 | 6 | 6 | 8 | 7 | 6 | 45

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Time Frame: From day 1 up to 4 months for participants assigned to the 0.03 or 0.1 mg/kg dose cohorts, up to 6 months for participants assigned to the 0.3 mg/kg dose cohort and for up to 9 months for participants assigned to the 1.0 or 3.0 mg/kg dose cohorts
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Denosumab 0.03 mg/kg | Denosumab 0.1 mg/kg | Denosumab 0.3 mg/kg | Denosumab 1.0 mg/kg | Denosumab 3.0 mg/kg
Number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 6
Participants
  Any adverse event | 6 | 2 | 3 | 5 | 6 | 5
  Serious adverse events | 0 | 0 | 0 | 0 | 0 | 0
  Treatment-related adverse events | 4 | 0 | 1 | 3 | 4 | 4
  Discontinuation due to adverse events | 0 | 0 | 0 | 0 | 0 | 0
  Deaths on study | 0 | 0 | 0 | 0 | 0 | 0

2. Secondary Outcome: Area Under the Serum Concentration Time Curve From Time 0 to Time of Last Quantifiable Serum Concentration (AUC0-t) of Denosumab
Time Frame: Day 1 predose and 5 minutes, 1, 4, 8, 12, 24, hours, days 3, 4, 5, 6, 8, 11, 15, 22, 29, 43, 57, 71, 85, 99, 113, also days 141 and 169 for participants in the 0.3, 1.0, or 3.0 mg/kg cohorts and days 197, 225, and 253 for the 1.0 or 3.0 mg/kg dose cohorts
Population: All participants who received denosumab
Measure: Mean (Standard Deviation); unit: μg*day/mL
Arm/Group | Denosumab 0.03 mg/kg | Denosumab 0.1 mg/kg | Denosumab 0.3 mg/kg | Denosumab 1.0 mg/kg | Denosumab 3.0 mg/kg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
μg*day/mL | 2.06 (0.53) | 15.2 (6.7) | 84.3 (20.1) | 481 (131) | 1790 (650)

3. Secondary Outcome: Maximum Observed Concentration of Denosumab (Cmax)
Time Frame: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Denosumab 0.03 mg/kg | Denosumab 0.1 mg/kg | Denosumab 0.3 mg/kg | Denosumab 1.0 mg/kg | Denosumab 3.0 mg/kg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
ng/mL | 99.6 (25.8) | 492 (166) | 1910 (658) | 8690 (2170) | 27400 (7880)

4. Secondary Outcome: Time to Maximum Observed Concentration (Tmax) of Denosumab
Time Frame: as for outcome 2
Population: All participants who received denosumab
Measure: Median (Full Range); unit: days
Arm/Group | Denosumab 0.03 mg/kg | Denosumab 0.1 mg/kg | Denosumab 0.3 mg/kg | Denosumab 1.0 mg/kg | Denosumab 3.0 mg/kg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
days | 7.0 [7 to 10] | 12.0 [7 to 21] | 14.0 [7 to 21] | 14.0 [10 to 21] | 14.0 [14 to 42]

5. Secondary Outcome: Apparent Clearance (CL/F) of Denosumab
Time Frame: as for outcome 2
Population: All participants who received denosumab
Measure: Mean (Standard Deviation); unit: mL/day/kg
Arm/Group | Denosumab 0.03 mg/kg | Denosumab 0.1 mg/kg | Denosumab 0.3 mg/kg | Denosumab 1.0 mg/kg | Denosumab 3.0 mg/kg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
mL/day/kg | 15.3 (4.2) | 8.31 (4.97) | 3.72 (0.89) | 2.20 (0.56) | 1.85 (0.58)

6. Secondary Outcome: Mean Residence Time (MRT) From Time 0 to Time of Last Quantifiable Serum Concentration
Time Frame: as for outcome 2
Population: All participants who received denosumab
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Denosumab 0.03 mg/kg | Denosumab 0.1 mg/kg | Denosumab 0.3 mg/kg | Denosumab 1.0 mg/kg | Denosumab 3.0 mg/kg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
days | 15.5 (4.7) | 22.5 (3.9) | 33.6 (5.8) | 42.6 (7.0) | 51.4 (5.8)

7. Secondary Outcome: Percent Change From Baseline in Urinary N-Telopeptide Corrected for Urine Creatinine (N-Tx/Cr)
Time Frame: Baseline and day 2, 3, 4, 5, 6, 8, 11, 15, 22, 29, 43, 57, 71, 85, 99, 113 (for all dose cohorts), 141, 169 (0.3, 1.0, and 3.0 mg/kg cohorts only), 197, 225, 253, 281, and 309 (1.0 and 3.0 mg/kg cohorts only).
Population: Treated participants with available data at each time point
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Denosumab 0.03 mg/kg | Denosumab 0.1 mg/kg | Denosumab 0.3 mg/kg | Denosumab 1.0 mg/kg | Denosumab 3.0 mg/kg
Number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 6
percent change
  Day 2 | 12 (11) | 6 (4) | -25 (8) | -22 (11) | -40 (7) | -64 (4)
  Day 3 | 19 (5) | -6 (7) | -30 (5) | -40 (11) | -51 (8) | -60 (3)
  Day 4 | 7 (6) | -18 (9) | -37 (16) | -48 (11) | -55 (6) | -62 (5)
  Day 5 | 23 (10) | -12 (12) | -44 (5) | -51 (8) | -53 (8) | -66 (6)
  Day 6 | 9 (7) | -1 (18) | -53 (8) | -62 (7) | -59 (6) | -72 (4)
  Day 8 | 16 (7) | -12 (13) | -55 (7) | -64 (5) | -57 (7) | -64 (10)
  Day 11 | 3 (8) | -36 (5) | -67 (5) | -65 (7) | -69 (6) | -79 (3)
  Day 15 | 4 (3) | -51 (4) | -68 (4) | -71 (5) | -71 (5) | -77 (5)
  Day 22 | -1 (5) | -41 (4) | -71 (6) | -70 (7) | -70 (5) | -82 (3)
  Day 29 | -1 (5) | -39 (5) | -68 (3) | -67 (6) | -64 (7) | -77 (4)
  Day 43 | -1 (5) | -33 (6) | -67 (4) | -68 (7) | -69 (8) | -81 (4)
  Day 57 | 0 (8) | -14 (3) | -59 (6) | -64 (8) | -56 (10) | -79 (6)
  Day 71 | -5 (7) | -23 (6) | -48 (10) | -65 (6) | -68 (5) | -82 (3)
  Day 85 | 8 (7) | 4 (8) | -48 (12) | -58 (9) | -68 (4) | -83 (4)
  Day 99 | 1 (6) | 4 (6) | -37 (15) | -64 (5) | -72 (4) | -77 (10)
  Day 113 | -5 (6) | 3 (4) | -30 (15) | -53 (10) | -77 (3) | -84 (2)
  Day 141: number analyzed (Participants) | 6 | 0 | 0 | 6 | 6 | 6
  Day 141 | -7 (9) |  |  | -51 (5) | -62 (5) | -81 (3)
  Day 169: number analyzed (Participants) | 6 | 0 | 6 | 6 | 6 | 6
  Day 169 | -15 (6) |  | 6 (14) | -41 (11) | -48 (9) | -78 (5)
  Day 197: number analyzed (Participants) | 4 | 0 | 0 | 0 | 6 | 6
  Day 197 | -3 (5) |  |  |  | -47 (8) | -79 (4)
  Day 225: number analyzed (Participants) | 5 | 0 | 1 | 5 | 6 | 6
  Day 225 | -7 (11) |  | 42.0 | -30 (4) | -20 (17) | -70 (4)
  Day 253: number analyzed (Participants) | 4 | 0 | 0 | 0 | 6 | 6
  Day 253 | -13 (10) |  |  |  | -25 (14) | -62 (5)
  Day 281: number analyzed (Participants) | 0 | 0 | 0 | 4 | 0 | 0
  Day 281 |  |  |  | -13 (8) |  |
  Day 309: number analyzed (Participants) | 0 | 0 | 0 | 0 | 4 | 6
  Day 309 |  |  |  |  | -19 (13) | -23 (12)

8. Secondary Outcome: Percent Change From Baseline in Bone-Specific Alkaline Phosphatase (BSAP)
Time Frame: Baseline and day 8, 15, 22, 29, 43, 57, 71, 85, 99, 113 (for all dose cohorts), 141, 169 (0.3, 1.0, and 3.0 mg/kg cohorts only), 197, 225, and 253, 281, and 309 (1.0 and 3.0 mg/kg cohorts only)
Population: Treated participants with available data at each time point
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Denosumab 0.03 mg/kg | Denosumab 0.1 mg/kg | Denosumab 0.3 mg/kg | Denosumab 1.0 mg/kg | Denosumab 3.0 mg/kg
Number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 6
percent change
  Day 8 | -0.4 (2.8) | -6.9 (5.9) | 16.6 (4.7) | 7.1 (2.0) | -0.5 (5.1) | 3.1 (6.4)
  Day 15 | -2.1 (1.4) | 1.1 (3.1) | 8.6 (2.0) | 13.2 (2.0) | 5.6 (5.9) | 11.5 (7.8)
  Day 22 | 1.1 (2.8) | 12.7 (3.1) | 5.8 (2.3) | 7.8 (3.8) | 7.0 (5.3) | 9.7 (5.8)
  Day 29 | 5.3 (2.9) | 8.9 (3.6) | 11.0 (3.5) | -0.7 (2.8) | 5.8 (4.2) | -0.4 (4.5)
  Day 43 | 3.6 (3.1) | -2.3 (2.8) | -7.6 (4.3) | -20.3 (3.2) | -10.2 (4.0) | -14.7 (2.6)
  Day 57 | 2.7 (1.6) | -5.9 (5.1) | -19.2 (2.8) | -33.1 (3.1) | -21.0 (4.9) | -24.0 (2.6)
  Day 71 | -0.9 (3.0) | -5.5 (4.8) | -29.0 (5.7) | -41.0 (2.2) | -36.1 (5.2) | -33.9 (4.7)
  Day 85 | 1.3 (2.2) | -7.9 (6.3) | -27.2 (6.1) | -47.7 (3.2) | -42.1 (4.2) | -43.9 (1.9)
  Day 99 | 1.7 (3.2) | -13.1 (3.3) | -33.4 (5.5) | -49.4 (3.0) | -44.0 (5.5) | -47.5 (2.7)
  Day 113 | 3.1 (2.3) | -0.5 (7.1) | -32.6 (5.4) | -54.2 (2.6) | -49.7 (5.1) | -51.4 (2.6)
  Day 141: number analyzed (Participants) | 6 | 0 | 0 | 6 | 6 | 6
  Day 141 | -0.2 (4.9) |  |  | -57.2 (2.6) | -50.7 (6.9) | -52.9 (3.8)
  Day 169: number analyzed (Participants) | 6 | 0 | 6 | 6 | 6 | 6
  Day 169 | 3.1 (4.3) |  | -33.9 (7.8) | -52.9 (2.5) | -50.1 (4.6) | -53.7 (2.9)
  Day 197: number analyzed (Participants) | 4 | 0 | 0 | 0 | 6 | 6
  Day 197 | 8.6 (5.8) |  |  |  | -43.9 (8.6) | -52.5 (2.7)
  Day 225: number analyzed (Participants) | 5 | 0 | 1 | 5 | 6 | 6
  Day 225 | 4.6 (3.0) |  | 19.5 | -37.1 (4.4) | -35.1 (8.5) | -48.4 (3.6)
  Day 253: number analyzed (Participants) | 4 | 0 | 0 | 0 | 6 | 6
  Day 253 | 11.7 (6.5) |  |  |  | -31.9 (9.7) | -44.0 (4.1)
  Day 281: number analyzed (Participants) | 0 | 0 | 0 | 4 | 0 | 0
  Day 281 |  |  |  | -10.7 (6.1) |  |
  Day 309: number analyzed (Participants) | 0 | 0 | 0 | 0 | 4 | 6
  Day 309 |  |  |  |  | -21.0 (14.7) | -26.8 (4.8)

9. Secondary Outcome: Percent Change From Baseline in Intact Parathyroid Hormone (iPTH)
Time Frame: Baseline and day 2, 3, 5, 8, 15, 29, 57, 85, 99, 113 (for all dose cohorts), 141, 169 (0.3, 1.0, and 3.0 mg/kg cohorts only), 197, 225, 253, 281, and 309 (1.0 and 3.0 mg/kg cohorts only)
Population: Treated participants with available data at each time point
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Denosumab 0.03 mg/kg | Denosumab 0.1 mg/kg | Denosumab 0.3 mg/kg | Denosumab 1.0 mg/kg | Denosumab 3.0 mg/kg
Number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 6
percent change
  Day 2 | 6.9 (8.7) | 2.4 (13.0) | 10.1 (14.1) | 44.0 (13.0) | 40.9 (19.5) | 129.0 (25.2)
  Day 3 | -8.2 (6.1) | 28.9 (9.7) | 15.0 (18.8) | 71.7 (15.8) | 60.7 (21.7) | 146.1 (46.0)
  Day 5 | -3.9 (6.0) | 47.6 (12.2) | 51.8 (17.9) | 114.2 (27.2) | 103.1 (41.8) | 262.1 (61.9)
  Day 8 | -0.7 (8.9) | 37.7 (20.4) | 76.9 (20.7) | 182.4 (40.2) | 163.7 (38.4) | 353.6 (92.4)
  Day 15 | 11.2 (8.9) | 91.5 (8.2) | 117.3 (33.4) | 146.4 (29.0) | 109.4 (36.3) | 203.2 (27.2)
  Day 29 | 5.1 (7.7) | 97.2 (23.8) | 110.9 (40.7) | 99.2 (16.8) | 70.4 (28.3) | 215.2 (79.4)
  Day 57 | 5.3 (8.3) | 64.6 (18.4) | 120.5 (35.5) | 98.0 (17.9) | 90.9 (20.8) | 177.0 (36.8)
  Day 85 | 17.1 (10.2) | 11.9 (9.6) | 36.6 (24.5) | 76.9 (20.2) | 64.4 (18.4) | 170.5 (40.8)
  Day 99 | 5.6 (7.4) | 19.9 (10.5) | 46.4 (31.1) | 79.6 (13.9) | 44.0 (10.9) | 178.5 (93.3)
  Day 113 | -1.2 (10.2) | 3.9 (15.4) | 29.5 (32.8) | 38.5 (13.5) | 46.5 (10.5) | 155.7 (44.5)
  Day 141: number analyzed (Participants) | 6 | 0 | 0 | 6 | 6 | 6
  Day 141 | -3.8 (13.9) |  |  | 16.9 (11.1) | 22.8 (16.6) | 175.4 (81.3)
  Day 169: number analyzed (Participants) | 6 | 0 | 6 | 6 | 6 | 6
  Day 169 | -7.9 (5.3) |  | -16.7 (10.6) | 19.7 (8.2) | 21.9 (16.1) | 90.2 (27.6)
  Day 197: number analyzed (Participants) | 4 | 0 | 0 | 0 | 6 | 6
  Day 197 | -14.9 (5.4) |  |  |  | 17.0 (9.8) | 100.7 (42.1)
  Day 225: number analyzed (Participants) | 5 | 0 | 1 | 5 | 6 | 6
  Day 225 | -5.1 (14.1) |  | 15.9 | -30.9 (5.0) | 6.2 (12.3) | 151.4 (83.5)
  Day 253: number analyzed (Participants) | 4 | 0 | 0 | 0 | 6 | 6
  Day 253 | 8.5 (12.6) |  |  |  | 10.9 (18.1) | 70.8 (31.5)
  Day 281: number analyzed (Participants) | 0 | 0 | 0 | 4 | 0 | 0
  Day 281 |  |  |  | -26.1 (9.4) |  |
  Day 309: number analyzed (Participants) | 0 | 0 | 0 | 0 | 4 | 6
  Day 309 |  |  |  |  | 16.6 (24.9) | 33.8 (11.9)

ADVERSE EVENTS:
Time Frame: From day 1 up to 4 months for participants assigned to the 0.03 or 0.1 mg/kg dose cohorts, up to 6 months for participants assigned to the 0.3 mg/kg dose cohort and for up to 9 months for participants assigned to the 1.0 or 3.0 mg/kg dose cohorts.
Description: Other Adverse Events summarizes the non-serious occurrences of adverse events that exceed the indicated frequency threshold.
Groups:
- Denosumab Total: All participants received a single subcutaneous injection of denosumab on day 1.
Arm/Group | Placebo | Denosumab 0.03 mg/kg | Denosumab 0.1 mg/kg | Denosumab 0.3 mg/kg | Denosumab 1.0 mg/kg | Denosumab 3.0 mg/kg | Denosumab Total
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/30
Other Adverse Events (participants affected / at risk) | 6/10 | 2/6 | 3/6 | 5/6 | 6/6 | 5/6 | 21/30
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=10) | Denosumab 0.03 mg/kg (N=6) | Denosumab 0.1 mg/kg (N=6) | Denosumab 0.3 mg/kg (N=6) | Denosumab 1.0 mg/kg (N=6) | Denosumab 3.0 mg/kg (N=6) | Denosumab Total (N=30)
ATRIAL FIBRILLATION (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
SENSATION OF BLOCK IN EAR (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
TINNITUS (Ear and labyrinth disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 1
BLEPHAROSPASM (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
CONJUNCTIVAL HAEMORRHAGE (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
CONJUNCTIVITIS (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 2
CHEILITIS (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
DIARRHOEA (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
GASTRITIS (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
GINGIVAL BLEEDING (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
LIP BLISTER (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
STOMACH DISCOMFORT (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
STOMATITIS (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 2
CHEST DISCOMFORT (General disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 2
CHEST PAIN (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
FATIGUE (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
INJECTION SITE ERYTHEMA (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
INJECTION SITE HAEMORRHAGE (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
INJECTION SITE PAIN (General disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 3
MALAISE (General disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 2
SEASONAL ALLERGY (Immune system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
BRONCHITIS ACUTE (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 1
HERPES ZOSTER (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 1
NASOPHARYNGITIS (Infections and infestations) | 3 | 1 | 2 | 0 | 5 | 1 | 9
PERIODONTAL INFECTION (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 1
BLISTER (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 1
CONTUSION (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 0 | 0 | 1
THERMAL BURN (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 1 | 2
HEPATIC ENZYME INCREASED (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 1 | 0 | 2
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 2
MUSCLE FATIGUE (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 1
MYALGIA (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
PERIARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
SPONDYLOSIS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
DIZZINESS (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
HEADACHE (Nervous system disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 2
HYPOAESTHESIA (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
RHINITIS ALLERGIC (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 2 | 0 | 3
DERMATITIS (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
DERMATITIS CONTACT (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
ECZEMA (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 2
HAEMORRHAGE SUBCUTANEOUS (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
PRURITUS (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
RASH (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.